CLINICAL TRIAL: NCT04286724
Title: Tackling Intrusive Traumatic Memories After a Difficult Birth: a proof-of Principle Study
Brief Title: Tackling Intrusive Traumatic Memories After a Difficult Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antje Horsch (Other)
Responsible Party: Sponsor-Investigator, Antje Horsch, Assistant Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01435
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Posttraumatic Stress Disorder; Intrusive Traumatic Memories
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single group pre-post study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Brief behavioural procedure including a computerized visuospatial task (computer game "Tetris")

INTERVENTIONS:
Behavioral: Brief behavioural procedure including a computerized visuospatial task (computer game "Tetris") — Brief behavioural procedure including a computerized visuospatial task (the computer game "Tetris") preceded by a reactivation of the traumatic memory of childbirth

SUMMARY:
This proof-of-principle study aims to investigate the effects of a brief behavioural procedure including a computerized visuospatial task (the computer game "Tetris") preceded by a reactivation of the traumatic memory of childbirth, on birth-related intrusive traumatic memories and other postpartum posttraumatic stress symptoms. Women who report birth-related intrusive memories after 6 weeks postpartum will monitor their intrusive traumatic memories in a daily diary. After two weeks of diary, they will meet a psychologist to briefly evoke the memory of their birth, and receive a brief behavioural procedure including playing Tetris. Participants will then continue to complete an intrusive traumatic memory diary during two weeks. It is predicted that they will report fewer intrusive memories in the two weeks following the intervention, compared to the two weeks before. This will inform the potential future development of a simple computerized intervention procedure to reduce distressing psychological symptoms after traumatic childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Gave birth at the Lausanne University Hospital
* Gave written consent
* Have at least 4 related-to-childbirth intrusions over the two weeks prior to recruitment, and at least 2 related-to-childbirth intrusions during the pre-intervention diary
* Gave birth more than 6 weeks ago
* Is able to distinguish intrusions linked to the traumatic childbirth from intrusions linked to other traumatic events

Exclusion Criteria:

* Gave birth to a stillborn child
* Not fluent in French
* Severe illness of mother or infant (e.g. cancer, cardiovascular disease, severe neurodevelopmental difficulties, malformations)
* Have an established intellectual disability, or psychiatric history such as psychotic illness
* Alcohol abuse and/or illegal drug use
* Currently receiving psychological care in relation with the traumatic birth experience

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Frequency of intrusive memories of the index trauma | Within 2 weeks following the intervention
  Frequency of intrusive traumatic memories related to childbirth recorded by participants in a trauma-related intrusive memories diary over the two weeks after the intervention

SECONDARY OUTCOMES:
Presence and severity of maternal PTSD symptoms | 1 month after the intervention
  PTSD Checklist (PCL-5) for DSM-5
Frequency of intrusive memories of the index trauma | Between 4 and 6 weeks after the intervention
  Frequency of intrusive traumatic memories related to childbirth recorded by participants in a trauma-related intrusive memories diary between the 4th and 6th weeks following the intervention
Psychological distress related to intrusive memories of the index trauma | Within 2 weeks following the intervention
  Rating scale for psychological distress related to intrusive memories related to childbirth that are reported in an intrusive memories diary over the two weeks after the intervention. It is a SUDS (Subjective Units of Distress Scale) from 1 to 10 (1= No distress at all while having the intrusion ; 10 = Extreme distress while having the intrusion).

OTHER OUTCOMES:
Intervention acceptability | 1 month after the intervention
  10-point Likert scale (1= The intervention was not at all acceptable; 10 = The intervention was extremely acceptable).

CONTACTS AND LOCATIONS:
Overall Officials: Antje Horsch, PhD, Principal Investigator — University of Lausanne and Lausanne University Hospital
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided